CLINICAL TRIAL: NCT02642198
Title: Clinical Investigation for Non-invasive Blood Pressure Monitor Accuracy Validation Performed on Neonatal, Infants and Children up to 3 Years Old
Brief Title: Non-Invasive Blood Pressure Monitor Accuracy in Neonatal Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mortara Instrument (Industry)
Responsible Party: Sponsor
Other Study IDs: 900_OPBG_2015
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Non-invasive Blood Pressure
Keywords: NiBP

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Surveyor S12 and S19 patient monitor — Non-invasive blood pressure measurement
  Other Names: S12/S19

SUMMARY:
This study is being conducted to validate the accuracy of non-invasive blood pressure (NIBP) measurement technology from Mortara Instrument, Inc. (Milwaukee, Wisconsin, USA) and Zoe Medical, Inc. (Topsfield, Massachusetts, USA) in a neonatal, infants and children up to 3 years old patient population. The study is defined according to the International Standard "ANSI/AAMI/ISO 81060-2:2013, Non-invasive sphygmomanometers - Part 2: Clinical investigation of automated measurement type".

DETAILED DESCRIPTION:
The device under test is Mortara Instrument's Surveyor S12/S19 patient monitors ("Surveyor") incorporating neonatal NIBP technology. Specifically, NIBP measurements will be taken using a cuff on the patient's limb (exact location will be determined by clinician) using a variety of cuffs sized for neonates and pediatrics. The device utilizes oscillometric technology to obtain quickly and conveniently non-invasive blood pressure measurements. Results will be compared to invasive blood pressure measurements from patients already monitored with such sensors. The Device under Test will be calibrated and verified by a Mortara representative on site.

ELIGIBILITY:
Patient inclusion criteria

Before proceeding with the blood pressure non-invasive measurements detection, patients shall be examined and met the following stated criteria:

* Patients shall have already an invasive blood pressure monitoring (with catheter), this criteria applies only for Method 1.
* It shall be possible to perform multiple measurements of Non Invasive Blood pressure on one or more limbs with inflatable cuff.
* Patient with weight and age range according to the protocol requirements previously defined.
* Once the patient is identify a pre-screening activities is performed in order to assess any differences in the blood pressure. If the differences are minimal, according to the criteria described in the next section "Exclusion criteria", the patient can be included in the study group.

Exclusion criteria

* Patients with unstable clinical or cardiovascular conditions;
* Patients with circulatory problems which can results in different blood pressure values in the limbs;
* patients with heart disease which can results in blood pressure wave morphology abnormalities;
* patients where the difference of systolic blood pressure between two limbs is greater than 15 mm Hg or the difference of lateral diastolic blood pressure is greater than 10mmHg;
* Patients with arrhythmias.

Ages: 29 Days to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include a minimum of 25 patients for the Method 1 and 20 patient for the Method 2, male and female, with the following weight and age (as defined by date of birth to current date; not gestational age) ranges:
  * At least 3 patients < 1,000 g in weight.
  * At least 3 patients 1,000 g to 2,000 g in weight.
  * At least 3 patients > 2,000 g in weight.
  * At least 3 patients ≥ to 29 days and < 1 year of age.
  * At least 3 patients ≥ 1 year and < 3 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To study is the non-invasive blood pressure measurements accuracy validation performed with the Surveyor S12 / S19 monitor in pediatric, infants and children up to 3 years patients per ISO 81060-2: 2013 requirements. | 4 hours per patient
  To study the accuracy of non-invasive blood pressure measurements in neonatal patients

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù (OPBG), Rome, Italy
  - U.O. Neonatal Intensive Care Immature Pediatric Hospital Bambino Gesù - IRCCS, Rome

IPD SHARING:
Plan to Share IPD: Undecided